CLINICAL TRIAL: NCT03398005
Title: A Phase 3, Multi-center, Placebo-controlled, Randomized, Double-blind 26-week Study to Assess the Safety and Efficacy of CaPre® in Patients With Severe Hypertriglyceridemia.
Brief Title: A Phase 3 STudy of CaPRe In LOwering Very hiGh TriglYcerides (TRILOGY 1)
Acronym: TRILOGY 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grace Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACA-CAP-001
Record Dates: First submitted 2017-11-21; First posted 2018-01-12 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Hypertriglyceridemia
Keywords: Omega-3 Fatty acids; Triglycerides
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CaPre (Experimental)
  Interventions: Drug: CaPre
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CaPre — 4 x 1 g capsules administered orally once a day for 26 weeks
  Arms: CaPre
Drug: Placebo — 4 x 1 g capsules administered orally once a day for 26 weeks
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the efficacy of CaPre 4 g daily, compared to placebo, in lowering fasting triglyceride (TG) levels in patients with fasting TG levels ≥500 mg/dL and ≤1500 mg/dL (≥5.7 mmol/L and ≤17.0 mmol/L) after 12 weeks of treatment.

Approximately 615 subjects will be screened to obtain 245 randomized subjects following a 2.5:1 treatment allocation ratio (CaPre: placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥18 years of age.
2. Isolated hypertriglyceridemia, with triglycerides ≥500 mg/dL and <1500 mg/dL (≥5.7 mmol/L and <17.0 mmol/L) OR Mixed hyperlipidemia, with serum triglycerides ≥500 and <1500 mg/dL treated with a statin, CAI or PCSK9I inhibitor, alone or in combination, that has been stable for 6 weeks prior to randomization. If the subject is not being treated and not contraindicated, a statin and/or CAI treatment may be initiated at the discretion of the Investigator at time of screening.
3. Willingness to maintain current physical activity level and follow the NCEP-TLC diet throughout the study.
4. Be informed of the nature of the study and give written consent prior to any study procedure.

Exclusion Criteria:

1. Allergy or intolerance to OM3 fatty acids, OM3-acid ethyl esters, OM3 phospholipids, fish, shell fish, or any component of the study medication.
2. Known lipoprotein lipase impairment or deficiency, or apo CII deficiency.
3. Subjects with lysosomal acid lipase deficiency.
4. Body mass index greater than 45 kg/m2.
5. Subjects who are pregnant, lactating, and subjects of childbearing potential who are either planning to become pregnant or who are not using acceptable birth control methods during study participation. Subjects of childbearing potential are subjects who have experienced menarche and do not otherwise meet the criteria for subjects not of childbearing potential, defined as:

   * Subjects who have had surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation); or
   * Subjects who are postmenopausal, i.e., who have had a cessation of menses for at least 12 months without an alternative medical cause. A follicle stimulating hormone (FSH) test ≥40 mIU/mL may be used to confirm the post-menopausal state in women not using hormonal contraception or hormonal replacement therapy.

   Subjects of childbearing potential must test negative for pregnancy at the time of enrollment and agree to use an acceptable contraceptive method or remain abstinent during the study or for at least 8 weeks following the last dose of study medication, whichever is longer.
6. Subjects taking tamoxifen, estrogens, or progestins, or other medications or nutritional supplements with mechanisms modifying estrogen or progestogen pathways, who have had dosage changes within 4 weeks prior to Visit 1.
7. Use of oral or injected corticosteroids or anabolic steroids within 6 weeks prior to randomization.
8. History of pancreatitis within the last 6 months prior to Visit 1.
9. History of symptomatic gallstone disease within the last 5 years, unless treated with cholecystectomy.
10. Diabetics requiring changes in medical therapy (other than short acting insulin dosage adjustments) within 6 weeks prior to Visit 1 or who have HbA1c greater than 9.5% at Visit 1.
11. Clinical or biochemical evidence of hyperthyroidism not stable with medication for at least 6 weeks prior to Visit 1.
12. Uncontrolled hypothyroidism or thyroid stimulating hormone (TSH) level more than 1.5 × upper limit of normal (ULN).
13. Thyroid hormone replacement therapy that has not been stable for more than 6 weeks prior to Visit 1.
14. History of cancer (other than basal cell carcinoma) within 2 years prior to Visit 1.
15. Cardiovascular event (i.e., myocardial infarction, acute coronary syndrome, new onset angina, stroke, transient ischemic attack, exacerbation of congestive heart failure requiring hospitalization or a change in treatment), life threatening arrhythmia, or revascularization procedure within 6 months prior to Visit 1.
16. Use of other prohibited drugs: weight loss prescription medications; human immunodeficiency virus (HIV) protease inhibitors; cyclophosphamide; isotretinoin; routine or anticipated use of systemic corticosteroids (local, topical, inhalation, or nasal corticosteroids are permitted); or anabolic steroids.
17. Use of any lipid-altering drug therapy, other than statins, CAI (such as ezetimibe) or PCSK9I inhibitors, alone or in combination, including niacin at a dose greater than 200 mg/day, fibrates, bile acid sequestrants, OM3 drugs (e.g., Lovaza or its generics,Vascepa, Epanova, Omtryg), OM3 supplements (e.g., fish oil, krill oil products), or any other herbal products or dietary supplements with potential lipid-altering effects. These products must be discontinued at least 6 weeks prior to randomization.
18. Resection of an aortic aneurysm or endovascular aortic repair within 6 months prior to Visit 1.
19. Recent history (within 6 months prior to Visit 1) or current significant nephrotic syndrome or ≥3 gram proteinuria daily, pulmonary, gastrointestinal, or immunologic disease.
20. Poorly controlled hypertension (systolic blood pressure ≥170 mmHg and/or diastolic blood pressure ≥100 mmHg). Subjects with hypertension adequately controlled with medication are eligible provided that their antihypertensive therapy has been stable for at least 4 weeks prior to Visit 1.
21. Recent history (past 12 months) of drug abuse or alcohol abuse, or alcohol use greater than 2 units per day (a unit of alcohol is defined as a 12-ounce (350 mL) beer, 5 ounce (150 mL) wine, or 1.5-ounce (45 mL) of 80-proof alcohol for drinks).
22. Hepatobiliary disease or serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5× ULN; if ALT/AST is >3× ULN, the levels must have been stable for 3 months prior to Visit 1.
23. Severe renal disease as defined by less than 30 mL/min serum creatinine clearance calculated using the Cockcroft-Gault formula.
24. Significant coagulopathy as defined by a known hereditary deficiency of coagulation factors or platelet function or an unexplained elevation of the prothrombin time (PT) international normalized ratio (INR) of ≥1.5. Subjects using warfarin [Coumadin®] or heparin are allowed. Subjects receiving other anticoagulants dabigatran, rivaroxaban, or apixaban are allowed. Subjects receiving acetylsalicylic acid (ASA) alone or in combination with other anti platelet agents (e.g., clopidogrel, prasugrel, ticagrelor) are also allowed.
25. Unexplained creatine kinase concentration 3 × ULN.
26. Creatine kinase elevation owing to known hereditary or acquired muscle disease.
27. Exposure to any investigational product, within 4 weeks prior to Visit 1.
28. Presence of any other condition the Investigator believes would interfere with the subject's ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the subject at undue risk.
29. Any life-threatening disease expected to result in death within 2 years, require frequent hospitalizations, extensive surgery or changes in medications or diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Percent change in fasting TG levels from baseline (average of Week -2, -1, and 0) to Week 12 (average of Week 11 and 12) in patients with fasting TG levels ≥500 mg/dL and ≤1500 mg/dL (≥5.7 mmol/L and ≤17.0 mmol/L). | Week 12

SECONDARY OUTCOMES:
Percent change from baseline (average of Week -2, -1, and 0) to Week 12 (average of Week 11 and 12) in non-HDL-C. | Week 12
Percent change from baseline (Week -1 and 0) to Week 12 (average of Week 11 and 12) in VLDL-C (β-quantification). | Week 12
Percent change from baseline (average of Week -2, -1, and 0) to Week 12 (average of Week 11 and 12) in HDL-C. | Week 12
Percent change from baseline (average of Week -1 and 0) to Week 12 (average of Week 11 and 12) in LDL-C (β-quantification). | Week 12

OTHER OUTCOMES:
Percent change from baseline (average of Week -2, -1, and 0) to all measured visits other than Week 12 (Week 4, Week 18 and Week 26) in TG (persistence of the effect of CaPre on TG). | Week 4; Week 18; Week 24
Proportion of subjects with a fasting TG level below 500 mg/dL (<5.7 mmol/L) at Week 12 and at Week 26. | Week 12; Week 26
Percent change from baseline (average of Week -2, -1, and 0) to Week 12 (average of Week 11 and Week 12) and Week 26 in TC. | Week 12; Week 26
Percent change from baseline (average of Week -1 and 0) to Week 12 (average of Week 11 and 12) and to Week 26 in RLP-C. | Week 12; Week 26
Percent change from baseline (average of Week -1 and 0) to Week 26 in LDL-C (β-quantification) and VLDL-C (β-quantification). | Week 26
Percent change from baseline (average of Week -2, -1, and 0) to Week 26 in non-HDL-C and HDL-C. | Week 26
Percent change from baseline (Week 0) to Week 12 and to Week 26 in apo B, apo A1, apo B/apo A1 ratio, apo CIII and apo A5. | Week 12; Week 26
Percent change from baseline (Week 0) to Week 12 and to Week 26 in lipoprotein particles concentration and size (LDL, non-HDL, HDL, IDL and VLDL). | Week 12; Week 26
Percent change from baseline (Week 0) to Week 12 and to Week 26 in oxidized LDL. | Week 12; Week 26
Percent change from baseline (Week 0) to Week 12 and to Week 26 in fasting serum glucose, insulin and HbA1c. | Week 12; Week 26
Percent change from baseline (Week 0) to Week 12 and to Week 26 in HOMA-IR and HOMA-β. | Week 12; Week 26
Percent change from baseline (Week 0) to Week 12 and to Week 26 in hs-CRP and Lp-PLA2. | Week 12; Week 26
Change from baseline (Week 0) to Week 4, Week 12, Week 18 and to Week 26 in Total plasma EPA concentration and Total plasma DHA concentration. | Week 4; Week 12; Week 18; Week 26
Percent change from baseline (Week 0) to Week 4, Week 12, Week 18 and to Week 26 in Total plasma EPA concentration and Total plasma DHA concentration. | Week 4; Week 12; Week 18; Week 26
Change from baseline (Week 0) to Week 12 and to Week 26 in OM3 Index. | Week 12; Week 26
Percent change from baseline (Week 0) to Week 12 and to Week 26 in OM3 Index. | Week 12; Week 26
Change from baseline (Week 0) to Week 12 and to Week 26 in AA. | Week 12; Week 26
Percent change from baseline (Week 0) to Week 12 and to Week 26 in AA. | Week 12; Week 26
Change from baseline (Week 0) to Week 12 and to Week 26 in omega-6/omega-3 ratio. | Week 12; Week 26
Percent change from baseline (Week 0) to Week 12 and to Week 26 in omega-6/omega-3 ratio. | Week 12; Week 26
Change from baseline (Week 0) to Week 12 and to Week 26 in EPA/AA ratio. | Week 12; Week 26
Percent change from baseline (Week 0) to Week 12 and to Week 26 in EPA/AA ratio. | Week 12; Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Mozaffarian, MD, DrPH, Principal Investigator — Tufts Friedman School of Nutrition Science and Policy
Locations (60):
- United States (60):
  - Research site, Birmingham, Alabama
  - Research site, Tucson, Arizona
  - Research site, Conway, Arkansas
  - Research site, El Cajon, California
  - Research site, Fresno, California
  - Research site, Garden Grove, California
  - Research site, Lomita, California
  - Research site, Newport Beach, California
  - Research site, Tustin, California
  - Research site, Boca Raton, Florida
  - Research site, Clearwater, Florida
  - Research site, Fort Myers, Florida
  - Research site, Hialeah, Florida
  - Research site, Homestead, Florida
  - Research site, Jacksonville, Florida
  - Research site, Kendall, Florida
  - Research site, Lake Worth, Florida
  - Research site, Miami, Florida
  - Research site, Miami Springs, Florida
  - Research site, North Miami Beach, Florida
  - Research site, Orlando, Florida
  - Research site, Pembroke Pines, Florida
  - Research site, Tamarac, Florida
  - Research site, Tampa, Florida
  - Research site, Wellington, Florida
  - Research site, West Palm Beach, Florida
  - Research site, Atlanta, Georgia
  - Research site, Gainesville, Georgia
  - Research site, Savannah, Georgia
  - Research site, Snellville, Georgia
  - Research site, Sugar Hill, Georgia
  - Research site, Meridian, Idaho
  - Research site, Gurnee, Illinois
  - Research site, Anderson, Indiana
  - Research site, Louisville, Kentucky
  - Research site, Eunice, Louisiana
  - Research site, Cadillac, Michigan
  - Research site, Jackson, Mississippi
  - Research site, Olive Branch, Mississippi
  - Research site, St Louis, Missouri
  - Research site, Omaha, Nebraska
  - Research site, Greensboro, North Carolina
  - Research site, Mooresville, North Carolina
  - Research site, Canton, Ohio
  - Research site, Marion, Ohio
  - Research site, Maumee, Ohio
  - Research site, Norman, Oklahoma
  - Research site, Beaver, Pennsylvania
  - Research site, Spartanburg, South Carolina
  - Research site, Chattanooga, Tennessee
  - Research site, Memphis, Tennessee
  - Research site, Arlington, Texas
  - Research site, Houston, Texas
  - Research site, Lampasas, Texas
  - Research site, San Antonio, Texas
  - Research site, Salt Lake City, Utah
  - Research site, West Jordan, Utah
  - Research site, Danville, Virginia
  - Research site, Bellevue, Washington
  - Research site, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mozaffarian D, Maki KC, Bays HE, Aguilera F, Gould G, Hegele RA, Moriarty PM, Robinson JG, Shi P, Tur JF, Lapointe JF, Aziz S, Lemieux P; TRILOGY (Study of CaPre in Lowering Very High Triglycerides) investigators. Effectiveness of a Novel omega-3 Krill Oil Agent in Patients With Severe Hypertriglyceridemia: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jan 4;5(1):e2141898. doi: 10.1001/jamanetworkopen.2021.41898. PMID 34989797